CLINICAL TRIAL: NCT06650527
Title: Effect of Cognitive Empathy Training on Dementia Caregivers
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Emory University (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Principal Investigator, James K. Rilling, Professor, Emory University
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: STUDY00007266; 1R01AG087216-01 (NIH)
Record Dates: First submitted 2024-10-18; First posted 2024-10-21 (Actual); Last update posted 2025-08-17 (Actual); Status verified 2025-08

CONDITIONS: Caregivers of People Living With Dementia; Dementia
Keywords: Cognitive empathy; People Living With Dementia; Caregivers
MeSH Terms: conditions — Dementia | interventions — Lead; Magnetic Resonance Spectroscopy

STUDY DESIGN:
Intervention Model Description: Using a crossover design, caregivers will be randomized to either cognitive empathy training (n=59) or a control condition (n=59). Neuroimaging, questionnaire, and biomarker data will be collected before the 10-day training, immediately after the training, and six months after. At the 6 month visit, participants will cross over to the other treatment
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group 1: Empathy Training (Experimental): Participants will be randomly assigned to the empathy training or control condition for 6 months. During the first phase of the study, participants in Group 1 will receive the photo captioning intervention.
  At the 6-month time point, participants in Group 1 will crossover to control.
  Assessments will be collected at baseline, 10-day (immediate post-training), 6-month (crossover), 6-month and 10-day (immediate post-crossover) and 12-month (completion)
  Interventions: Behavioral: Cognitive Empathy Training; Procedure: Pre and post intervention blood spot collection; Procedure: Pre and post intervention MRI session
- Group 2: Control Condition (Other): During the first phase of the study, participants in Group 2 are controls. At the 6-month time point, participants in Group 2 will crossover and initiate the intervention.
  Assessments will be collected at baseline, 10-day (immediate post-training), 6-month (crossover), 6-month and 10-day (immediate post-crossover), and 12-month (completion)
  Interventions: Behavioral: Control Condition; Procedure: Pre and post intervention blood spot collection; Procedure: Pre and post intervention MRI session

INTERVENTIONS:
Behavioral: Cognitive Empathy Training — Participants will engage in a mentalization activity by captioning photos of their care recipients, reflecting on what the care recipient might be thinking or feeling. Over 10 days, caregivers will take 3-5 daily pictures of their care recipient and caption each with descriptive text representing the recipient's inner voice. This task encourages caregivers to consider the care recipient's perspective and motivations behind their behavior or emotional experiences. Photos will be shared securely via encrypted email. Utilizing accessible smartphone technology, the study allows caregivers to capture and reflect on meaningful moments with their care recipients
  Arms: Group 1: Empathy Training
Behavioral: Control Condition — In the control condition, participants will be asked to take 3-5 daily photographs of nature over 10 days. They will be asked to caption each photo with a description of what they see. This exercise will involve many of the same activities as the cognitive empathy training, except that participants will not be mentalizing or taking the the perspective of their PLWD or anyone else.
  Arms: Group 2: Control Condition
Procedure: Pre and post intervention blood spot collection — At their initial study visit, participants will provide a blood spot sample for measurement of C-reactive protein, pro-inflammatory cytokines and Epstein-Barr virus antibody titers.
  Other Names: Labs
Procedure: Pre and post intervention MRI session — In this study, caregivers will be positioned in a Siemens Trio 3T MRI scanner for functional imaging. They will view images of their care recipient care recipient, other similar care recipients care recipient, and photographs of friends or family members, pressing a button each time they see their care recipient care recipient's photo to monitor attention. The task involves viewing eight photos of four individuals with happy and neutral expressions, followed by rest periods. This sequence repeats five times, with each stimulus presented for 5 seconds and inter-trial intervals of 2, 3, or 4 seconds, totaling 11 minutes and 15 seconds. A subsequent 10-minute diffusion-weighted scan will assess brain white matter integrity, using 60 diffusion directions. All scans will be completed within 40 minutes.
  Other Names: MRI scan

SUMMARY:
The goal of this project is to investigate the effect of cognitive empathy training on mental health, inflammation, and immune function in caregivers of people living with dementia (PLWD), and to examine the underlying psychological and neurobiological mechanisms.

The primary aim is to establish the effectiveness of cognitive empathy training in improving caregiver mental health and immune function, and in decreasing caregiver inflammation

The secondary aim is to investigate the psychological and neurobiological mechanism by which cognitive empathy training improves caregiver well-being

DETAILED DESCRIPTION:
In the U.S., over 7 million people currently live with Alzheimer's disease and related disorders (ADRD), a number projected to exceed 16 million by 2060. Family caregivers, numbering more than 11 million, play a crucial role in managing the care of these individuals, often bearing significant emotional and financial burdens. In 2021, the cost of care for dementia reached $593 billion, with families contributing a substantial portion. Caregivers frequently experience negative mental and physical health impacts due to chronic stress, including increased rates of depression and inflammation. Research indicates that caregiving leads to decreased immune function, with elevated Epstein-Barr virus antibody titers serving as a marker for immune health. Interventions aimed at supporting caregivers, such as psychoeducational programs, have shown benefits, particularly in enhancing coping skills. Additionally, fostering cognitive empathy in caregivers may improve their mental health and the quality of care provided to individuals with dementia, potentially mitigating some of the adverse health effects associated with caregiving stress.

ELIGIBILITY:
Inclusion Criteria:

* Caregivers must live with their care recipient
* Caregivers must have a Zarit Burden Scale score of 19 or higher
* Caregivers must have no plans to move their care recipient to an institutional setting within the next year
* Caregivers must be able to read and write English
* Care recipient not in hospice
* Access to a mobile phone that can take and email photographs

Exclusion Criteria:

* Subjects with a history of seizures or other neurological disorders, alcoholism, or any other substance abuse
* Subjects with a history of psychiatric illness (excluding depression and anxiety disorders) will also be excluded
* Subjects with a history of head trauma based on Survey
* Subjects with MRI contra-indications

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 118 (Estimated)
Dates: Start 2025-02-13 (Actual); Primary Completion 2028-11-01 (Estimated); Study Completion 2028-11-01 (Estimated)

PRIMARY OUTCOMES:
Zarit Burden Scale score | Baseline, immediately post-training (10-Day) , 6 months post-training
  Zarit Burden Inventory (ZBI) score is a 22-item Likert scale. Each item is a statement which the caregiver is asked to endorse using a 5-point scale. Response options range from 0 (Never) to 4 (Nearly Always). Total score is obtained by summing all items endorsed. Higher scores indicate greater perceived burden.
The Center for Epidemiological Studies Depression (CESD) Scale score | Baseline, immediately post-training (10-Day), 6 months post-training
  The CESD-R is a 20 item Likert scale scored 0-3 with somatic and psychological subscales. Total scores range from 0 to 60, with high scores indicating greater depressive symptoms.
The State/Trait Anxiety Index (STAI) score | Baseline, immediately post-training (10-Day), 6 months post-training
  The STAI State (STAI-S) is a 20-item 4-point Likert scale commonly used measure of state anxiety. Respondents report the intensity of their anxiety at that moment on a 4-point scale where 1 = not at all and 4 = very much so. Total scores range from 20 to 80 and higher scores indicate greater anxiety.
Perspective-taking subscale if the Interpersonal Reactivity Index (IRI) | Baseline, immediately post-training (10-Day), 6 months post-training
  The Perspective-Taking scale of the IRI ranges from 0-28, and higher scores are a better outcome
Dyadic Relationship Scale score | Baseline, immediately post-training (10-Day), 6 months post-training
  The Dyadic Relationship Scale ranges from 0-33 and higher scores are a worse outcome.
IL-6 levels | Baseline, immediately post-training (10-Day), 6 months post-training
  Cytokine (Measure of inflammation)
IL-10 levels | Baseline, immediately post-training (10-Day), 6 months post-training
  Cytokine (Measure of inflammation)
TNF-α levels | Baseline, immediately post-training (10-Day), 6 months post-training
  Cytokine (Measure of inflammation)
Epstein-Barr virus antibody titers | Baseline, immediately post-training (10-Day), 6 months post-training
  Measure of immune system functioning
fMRI activation within dorsomedial prefrontal cortex (DMPFC) for contrast (own person - unknown person) | Baseline, immediately post-training (10-Day), 6 months post-training
  Measure of activation within one cognitive empathy ROI
fMRI activation within precuneus for contrast (own person - unknown person) | Baseline, immediately post-training (10-Day), 6 months post-training
  Measure of activation within one cognitive empathy ROI
fMRI activation within temporo-parietal junction for contrast (own person - unknown person) | Baseline, immediately post-training (10-Day), 6 months post-training
  Measure of activation within one cognitive empathy (region of interest) ROI
fMRI activation within ventrolateral prefrontal cortex for contrast (own person - unknown person) | Baseline, immediately post-training (10-Day), 6 months post-training
  Measure of activation within an emotion regulation ROI

CONTACTS AND LOCATIONS:
Overall Officials: James Rilling, PhD, Principal Investigator — Emory College of Arts & Sciences; Kenneth Hepburn, PhD, Principal Investigator — Emory School of Nursing
Locations (3):
- United States (3):
  - Alter, Atlanta, Georgia
  - Emory Integrated Memory Care, Atlanta, Georgia
  - NIA Goizueta Alzheimer's Disease Research Center, Atlanta, Georgia

IPD SHARING:
Plan to Share IPD: Yes
All behavioral, neuroimaging, and inflammation biomarker data will be preserved and shared. Photo captions will be shared without the photographs. In addition, basic participant demographics and ID numbers will be provided.
Supporting Information: Study Protocol, SAP
Time Frame: Data will be made available no later than the time of an associated publication or the end of the performance period, whichever comes first
Access Criteria: Open Science Framework